CLINICAL TRIAL: NCT04217343
Title: NON-COMPLEMENT MEDIATED AMR vs. COMPLEMENT MEDIATED AMR: DOES DD-cfDNA/GEP SHOW A DIFFERENCE
Brief Title: NCAMR-CAMR Allosure Study
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Tampa General Hospital (Other)
Responsible Party: Principal Investigator, Benjamin Mackie, Principal Investigator/Medical Doctor, Tampa General Hospital
Other Study IDs: 19-0118
Record Dates: First submitted 2019-12-09; First posted 2020-01-03 (Actual); Last update posted 2022-08-22 (Actual); Status verified 2022-08

CONDITIONS: Transplant Failure
Keywords: Heart

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- non-complement mediated pAMR(H+)
  Interventions: Diagnostic Test: Allosure/Allomap/Cytokines testing
- complement mediated pAMR(I+)
  Interventions: Diagnostic Test: Allosure/Allomap/Cytokines testing

INTERVENTIONS:
Diagnostic Test: Allosure/Allomap/Cytokines testing — All patients with evidence of Cardiac Transplant rejection will undergo Allosure, Allomap, and cytokine testing. Allosure and Allomap will be performed as part of routine care. Cytokine testing will be performed at time of rejection and resolution.

SUMMARY:
Heart Transplant recipients at Tampa General Hospital heart transplant program who have pAMR1(H+) or pAMR1(I+) rejection will have a DD-cfDNA /GEP sample obtained at the time of the rejection. The DD-cfDNA/GEP will then be drawn every month post treatment for the rejection until the DD-cfDNA/GEP level returns to normal. A total of fifteen recipients with pAMR1(H+) and fifteen recipients with pAMR1(I+) rejection will be included in the study which will last two years. The presence of HLA antibodies (DSA's) and the titers, presence of Autoantibodies, the measurement of cytokines IL2, IL4, IL6, IL 10, IL 17, TNF alpha, TGF beta, the presence of coronary artery vasculopathy, the time from transplant to the onset of the episode of AMR, time to resolution, the response to treatment and comparison to the DD-cfDNA/GEP level with pAMR2 and pAMR 3 rejections will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have undergone Orthotopic Heart Transplantation who have pAMR1 rejection.

Exclusion Criteria:

* Subjects less than 18 years old

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have undergone Orthotopic Heart Transplantation who have pAMR1 rejection will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2020-03-05 (Actual); Primary Completion 2023-03-05 (Estimated); Study Completion 2023-03-05 (Estimated)

PRIMARY OUTCOMES:
The level of dd-cfDNA in non-compliment mediated pAMR1 (H+) and complement mediated pAMR1 (I+) heart transplant rejection will be measured. | 2 years
  The level of dd-cfDNA in non-compliment mediated pAMR1 (H+) and complement mediated pAMR1 (I+) heart transplant rejection will be measured and then compared statistically to each other via Students t test as well as to the level of dd-cf DNA before and after the rejection episode.

SECONDARY OUTCOMES:
The level of inflammatory cytokines in non-compliment mediated pAMR1(H+) and compliment mediated pAMR1(I+) heart transplant rejection will be measured. | 2 years
  The level of inflammatory cytokines in non-compliment mediated pAMR1(H+) and compliment mediated pAMR1(I+) heart transplant rejection will be measured and compared statistically to each other via the Students t test as well as to the level of inflammatory cytokines after the rejection episode has resolved. The cytokines that will be assessed are: IL2, IL4, IL6, IL10, IL17, TNF alpha and TGF beta.
The presence of HLA antibodies (DSA's) and titer levels, autoantibodies and titer levels and coronary artery vasculopathy will be measured. | 2 years
  The presence of HLA antibodies (DSA's) and titer levels, autoantibodies and titer levels and coronary artery vasculopathy will be measured in the heart transplant recipients with non-compliment mediated pAMR1(H+) and pAMR1(I+) rejection and compared to each other via Students t test.

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Mackie, MD, Principal Investigator — Tampa General Hospital/Tampa General Medical Group
Locations (1):
- Tampa General Hospital, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: No